CLINICAL TRIAL: NCT02355080
Title: A Bundled Rapid HIV/HCV Testing Intervention to Increase Receipt of Test Results
Acronym: iKnow2 Project
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York University (Other); Beth Israel Medical Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jemima Frimpong, Assistant Professor of Health Policy and Management, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAN5869; R34DA038530 (NIH)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Substance-related Disorders
Keywords: HIV; HCV
MeSH Terms: conditions — Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-site bundled rapid HIV/HCV testing (Experimental): Participants will receive the on-site bundled rapid HIV/HCV testing intervention. In the intervention group, all patients will receive an offer to participate in rapid HIV/HCV testing. Those who accept this offer will: receive pre-test information about testing procedures and education, be tested, receive results during the same visit as testing, and be provided post-test counseling and support services by trained test counselors. Patients with a preliminary positive (i.e., reactive) HIV and/or HCV test result(s) will be actively linked immediately to a health care provider for further evaluation and confirmatory HIV and/or HCV RNA testing.
  Interventions: Behavioral: On-site bundled rapid HIV/HCV testing
- Standard of care (SOC) (Active Comparator): Participants will receive the standard of care (SOC) at the study sites. The SOC entails venipuncture whole blood HIV testing + venipuncture whole blood HCV testing. Blood draws are sent to an external laboratory for processing, and patients must return for test results in another visit. Patients may not receive pre-test information or results and post-test counseling, especially if non-reactive or negative test result(s). Reflex testing is not standard practice, therefore some patients may require another visit and blood draw for confirmatory HIV and/or HCV RNA testing. Linkage to care in the SOC is accomplished by referral to a health care provider, either within the participating substance use disorder treatment organization or passive referral to other health facilities.
  Interventions: Behavioral: Standard of care (SOC)

INTERVENTIONS:
Behavioral: On-site bundled rapid HIV/HCV testing — Participants will be offered bundled on-site rapid HIV and HCV testing with post-test counseling that addresses both sexual and drug use risk reduction, and linkage to care.
  Arms: On-site bundled rapid HIV/HCV testing
Behavioral: Standard of care (SOC) — Participants will receive the SOC for HIV and HCV testing at the study sites.
  Arms: Standard of care (SOC)

SUMMARY:
This is a randomized controlled clinical trial in which adults receiving drug abuse treatment will be recruited to participate in a HIV and hepatitis C (HCV) testing study. The purpose of this study is to test the efficacy of two HIV/HCV testing strategies on increasing receipt of test results: (1) on-site bundled rapid HIV/HCV testing (i.e., joint offer of HIV and HCV at the point of encounter), and (2) standard of care for HIV and HCV testing.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial in which adults receiving drug abuse treatment will be recruited to participate in a HIV and hepatitis C (HCV) testing study. The purpose of this study is to test the efficacy of two HIV/HCV testing strategies on increasing receipt of test results: (1) on-site bundled rapid HIV/HCV testing (i.e., joint offer of HIV and HCV at the point of encounter), and (2) standard of care for HIV and HCV testing. Secondary outcomes include linkage to care and HIV and HCV risk behaviors. Participants will complete a baseline assessment to report their demographics, sexual risk behaviors, drug-using risk behaviors, utilization of drug abuse treatment services and will be randomized to one of two groups. At one-month post-randomization, participants will complete a follow-up assessment to determine whether or not they received their HIV or HCV test results. At three months post-randomization, participants will complete a follow-up assessment to assess linkage to care and changes, if any, in their HIV and HCV sexual risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Report being HIV and HCV negative, or report not knowing HIV and HCV status
* Not have received results of an HIV or HCV test initiated within the last 12 months
* Able and willing to provide informed consent
* Seeking or currently receiving drug (excluding alcohol only treatment) abuse treatment services at the participating treatment programs
* At least 18 years old
* Able to communicate in English
* Willing to sign a release form that will allow medical record review (to corroborate self-reports of receipt of test results)
* Able and willing to provide locator information (contact number and address) for follow-up surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Self-Report Receipt of HIV and Hepatitis C Test Results | One month post-randomization
  The primary outcome is self-reported receipt of HIV/HCV test results. This will be measured at one-month post-randomization for all participants. We acknowledge that there are several potential HIV/HCV testing behaviors that could be evaluated in this study: acceptance of testing, completion of testing, and receipt of testing results, either HIV or HCV. Acceptance of testing measures whether or not a participant would accept the offer of an HIV or HCV test. Completion of testing measures whether or not a participant completes the HIV or HCV test. Receipt of test results refers to whether or not a participant self-reports having received the results of the HIV or HCV test.

SECONDARY OUTCOMES:
Linkage to care (Proportion of patients who initiated HIV/HCV care before the 3-month follow-up among those whose test results were positive for HIV and/or HCV.) | One month post-randomization
  Proportion of patients who initiated HIV/HCV care before the 3-month follow-up among those whose test results were positive for HIV and/or HCV.
Sexual risk behaviors (Counts of unprotected vaginal and anal sex acts in the past 3 months with any sex partner.) | One month post-randomization
  Counts of unprotected vaginal and anal sex acts in the past 3 months with any sex partner.
Drug use behaviors (Prevalence of use of any drugs in the past 3 months; and unsafe injection practices.) | One month post-randomization
  Prevalence of use of any drugs in the past 3 months; and unsafe injection practices.

CONTACTS AND LOCATIONS:
Overall Officials: Jemima A. Frimpong, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- Acacia Network/Promesa, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frimpong JA, D'Aunno T, Perlman DC, Strauss SM, Mallow A, Hernandez D, Schackman BR, Feaster DJ, Metsch LR. On-site bundled rapid HIV/HCV testing in substance use disorder treatment programs: study protocol for a hybrid design randomized controlled trial. Trials. 2016 Mar 3;17(1):117. doi: 10.1186/s13063-016-1225-4. PMID 26936623